CLINICAL TRIAL: NCT02116478
Title: Gastrocnemius Recession vs. Conservative Treatment for Chronic Plantar Fasciitis. A Randomized Controlled Trial.
Brief Title: Gastrocnemius Recession vs. Conservative Treatment for Chronic Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marius Molund, MD, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/2055
Record Dates: First submitted 2014-04-08; First posted 2014-04-17 (Estimated); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; gastrocnemius recession
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gastrocnemius recession (Experimental): gastrocnemius recession
  Interventions: Procedure: surgical proximal medial gastrocnemius recession

INTERVENTIONS:
Procedure: surgical proximal medial gastrocnemius recession — proximal medial gastrocnemius recession

SUMMARY:
The purpose of the study is to compare the clinical results for patients suffering from plantar fasciitis treated with gastrocnemius recession vs. conservative treatment.

DETAILED DESCRIPTION:
All patients will be instructed in stretching exercises. Half of the patients will be randomized to proximal medial gastrocnemius recession. All patients will be followed for 1 year. Additional long term follow-up will be 6 years after inclusion

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of plantar fasciitis lasting more than 12 months.
* Isolated gastrocnemius contracture

Exclusion Criteria:

* No previous surgery to foot or ankle
* No active arthritis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in American Orthopaedic foot and ankle society (AOFAS) ankle-hindfoot score | 1 year and 6 years postoperative
  The change in AOFAS from baseline to follow-up, as well as the difference between the groups treated non-operatively and operatively will be reported on a 0-100 scale.

SECONDARY OUTCOMES:
0-10 points Visual analog pain score | 1 year and 6 years postoperative
  Difference in pain between groups will be reported on 0-10 points visual analog scale

OTHER OUTCOMES:
Short form-36 (SF-36) | 1 year and 6 years postoperative
  Difference in subgroup parameters between baseline and follow-up as well as between group differences will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Marius Molund, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No